CLINICAL TRIAL: NCT06315647
Title: Comparative Study Between Double Guide Wire Technique Versus Trans Pancreatic Sphincterotomy Versus Precut and Fistulotomy Techniques for Difficult Biliary Cannulation
Brief Title: Comparison Between Different Techniques in Difficult CBD Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed El Said Salam, Dr, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Difficult CBD cannulation
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: ERCP, Difficult CBD Cannulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients enrolled for double guide wire technique. (Active Comparator)
  Interventions: Procedure: DGT vs TPS vs Precut and fistulotomy in Difficult CBD cannulation
- Patients enrolled for trans - pancreatic sphincterotomy technique. (Active Comparator)
  Interventions: Procedure: DGT vs TPS vs Precut and fistulotomy in Difficult CBD cannulation
- Patients enrolled for needle knife precut technique or fistulotomy technique. (Active Comparator)
  Interventions: Procedure: DGT vs TPS vs Precut and fistulotomy in Difficult CBD cannulation

INTERVENTIONS:
Procedure: DGT vs TPS vs Precut and fistulotomy in Difficult CBD cannulation — comparison between different technique in difficult CBD cannulation

SUMMARY:
This study aims to compare the efficacy and outcomes between double guidewire technique (DGT), trans pancreatic sphincterotomy (TPS) as well as precut and fistulotomy techniques in ERCP in patients defined as having difficult biliary cannulation.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is the standard procedure for diagnostic and therapeutic interventions for pancreatobiliary diseases. Bile duct cannulation is the most basic and important technique for carrying out diagnostic and therapeutic biliary interventions.

Since the advent of ERCP selective cannulation of the biliary duct is the most important step for successful treatment of biliary tract diseases during ERCP procedures, despite various accessory devices, the standard biliary cannulation technique has been reported to fail in approximately 5-20% cases.

Various endoscopic techniques for Selective Bile duct cannulation have been reported, including standard techniques (e.g. contrast injection technique, wire-guided cannulation ), pancreatic guidewire technique (e.g. double guidewire technique [DGW]), precut sphincterotomy, endoscopic papillectomy, endoscopic ultrasound-guided rendezvous procedure, and percutaneous transhepatic biliary drainage-guided procedure.

Bile duct cannulation can be difficult because of; different anatomical features, inflammatory processes, and adenomas of the papilla or periampullary diverticulum. Large prospective studies have demonstrated that difficult cannulation is an independent risk factor for post ERCP pancreatitis.

As the technique developed, several supplementary techniques have been recommended to facilitate the access to the common bile duct in cases of standard biliary cannulation failure, these are known to significantly increase not only the success rate of selective biliary cannulation but also the complication rate .

Commonly, a precutting technique is used to allow biliary access when the standard cannulation technique failed. There are types of precutting technique: needle-knife papillotomy, suprapapillary fistulotomy and trans pancreatic sphincterotomy, in terms of effectiveness and efficiency of the precutting technique, TPS, which does not need avoiding pancreatic duct cannulation unintentionally, is an effective method especially for difficult biliary cannulation.

Also, the use of a guidewire to physically occupy the pancreatic duct, also known as the double guidewire technique, this method has been used with promising results in cases of complex biliary cannulation, especially in patients with a distorted BD anatomy caused by neoplasia or atypical morphology of the ampulla.

ELIGIBILITY:
Inclusion Criteria:

* Patients having different biliary tract disorders for which ERCP is indicated and after which they defined as having difficult CBD cannulation.

Exclusion Criteria:

1. Age of less than18 years.
2. Coagulopathy in terms of INR>2.
3. Patients with severe heart disease defined as patients with decompensated heart diseases or EF > 40%.
4. Subjects who underwent prior biliary or pancreatic sphincterotomy or dilatation or stenting of either duct.
5. Complicated acute pancreatitis defined as patients with moderate to sever acute pancreatitis according to Revised ATLANTA criteria 2012.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Comparative Study Between Different Interventional Techniques for Difficult Common Bile Duct Cannulation In Endoscopic Retrograde Cholangio-pancreatography | Baseline
  compare efficacy of different cannulation techniques for difficult CBD cannulation

CONTACTS AND LOCATIONS:
Locations (1):
- National liver Institute, Shibīn al Kawm, Menofia, Egypt

REFERENCES:
- [Background] Miao L, Li QP, Zhu MH, Ge XX, Yu H, Wang F, Ji GZ. Endoscopic transpancreatic septotomy as a precutting technique for difficult bile duct cannulation. World J Gastroenterol. 2015 Apr 7;21(13):3978-82. doi: 10.3748/wjg.v21.i13.3978. PMID 25852284
- [Background] Yoo YW, Cha SW, Lee WC, Kim SH, Kim A, Cho YD. Double guidewire technique vs transpancreatic precut sphincterotomy in difficult biliary cannulation. World J Gastroenterol. 2013 Jan 7;19(1):108-14. doi: 10.3748/wjg.v19.i1.108. PMID 23326171
- [Background] Huang L, Yu QS, Zhang Q, Liu JD, Wang Z. Comparison between double-guidewire technique and transpancreatic sphincterotomy technique for difficult biliary cannulation. Dig Endosc. 2015 Mar;27(3):381-7. doi: 10.1111/den.12387. Epub 2014 Nov 11. PMID 25284147